CLINICAL TRIAL: NCT05997316
Title: Assessing the Feasibility and Acceptability of a Time Restricted Feeding Intervention Among Older Adults With Mild Cognitive Impairment
Brief Title: Time Restricted Eating for Metabolic and Psychological Optimization
Acronym: TEMPO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Duke University (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-2774; 1R61AG080615-01 (NIH)
Record Dates: First submitted 2023-08-10; First posted 2023-08-18 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Mild Cognitive Impairment; Obesity
MeSH Terms: conditions — Cognitive Dysfunction; Obesity

STUDY DESIGN:
Masking Description: Assessors will be blinded to the participant's intervention fidelity and engagement.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Time restricted eating (Experimental): Participants will engage in a 12-week time restricted fasting intervention. Each week, participants will work with a clinical psychologist to modify the timing of their eating behaviors to adhere to a 16-hour fast, 2-3 days per week.
  Interventions: Behavioral: Time restricted eating

INTERVENTIONS:
Behavioral: Time restricted eating — Participants will work with a psychologist towards achieving a 16 hour fasting period, 2-3 days per week. The intervention will last 12 weeks, with different intervention materials gradually introduced over the course of the 12 weeks.

SUMMARY:
Obesity and related metabolic comorbidities have been associated with more than a 4-fold increased risk of incident cognitive impairment, including Alzheimer's disease and related dementias (ADRD). Dysfunctional metabolic flexibility is increasingly recognized as a critical mechanism linking metabolic risk factors to risk of cognitive impairment, although few studies portable behavioral strategies to enhance metabolic function among individuals at risk for ADRD. The present study will examine the feasibility and acceptability of a 12-week time restricted feeding intervention among individuals with mild cognitive impairment (MCI). Changes in cognitive and metabolic function will also be examined.

DETAILED DESCRIPTION:
Obese older adults with mild cognitive impairment with mild cognitive impairment will be asked to participate in a 12 week time restricted fasting intervention. Working with a behavioral psychologist, they will adapt the timing their eating patterns to incorporate 2-3 days per week with a 16 hour fasting period, typically lasting from after dinner to lunch the next day. The behavioral intervention will titrate fasting using established behavioral change techniques, with early phase sessions focusing on organizational principles to prepare for weekly fasting scheduling and acceptance-based psychological coping skills, including the ability to tolerate symptoms of hunger and discomfort that may accompany fasting. After treatment initiation, sessions will focus on broadening fasting behaviors for flexible adoption across different contexts and to enhance maintenance of fasting patterns. At baseline and following treatment, participants will undergo tests of cognitive and metabolic function to assess memory, executive function, metabolic flexibility, and inflammation. At both time points, participants will also undergo an abbreviated assessment of cognitive and metabolic function under fasting conditions to assess for any cognitive weaknesses unmasked during periods of brief metabolic 'stress'.

ELIGIBILITY:
Inclusion Criteria:

Subjects will include those men and women:

* aged 65-80 years,
* with amnestic Mild Cognitive Impairment (Montreal Cognitive Assessment Battery score [MoCA] total score 19-25; and score of > 1.0 on the Mail-in Cognitive Function Screening Instrument),
* obese (body mass index 30-40 kg/m^2),
* sedentary, and
* willing to participate in all aspects of the proposed intervention.

Exclusion Criteria:

Reasons for participant exclusion will include:

* secondary causes of obesity,
* evidence of clinical dementia (MoCA score < 18), severe chronic kidney disease (eGFR <45 ml/min/1.73m^2),
* heart failure,
* high grade arrhythmias,
* severe valvular heart disease,
* severe asthma or chronic obstructive lung disease,
* diabetes requiring insulin,
* musculoskeletal or neurologic problems that would preclude participation in aerobic exercise training,
* a major psychiatric disorder,
* a history of drug abuse,
* alcohol consumption >14 drinks/week,
* gastric bypass surgery,
* non-English speaking, or
* a life-limiting comorbid medical condition (e.g. cancer).

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 33 (Actual)
Dates: Start 2023-08-07 (Actual); Primary Completion 2025-06-26 (Actual); Study Completion 2025-06-26 (Actual)

PRIMARY OUTCOMES:
Memory | Baseline and 12 Weeks
  The primary Memory outcome measure will be a mean-rank, global score comprised of the following subtests. The Hopkins Verbal Learning Test Revised will assess verbal memory on a list learning task. Scores range from 0 to 12 across three learning trials with higher scores indicating better performance. A total learning score therefore ranges from 0 to 36 and a delayed memory score of 0 to 12, with higher scores reflecting better performance. The Brief Visual Memory Test - Revised will be used to assess visual learning and memory. Scores range from 0 to 12 across three learning trials with higher scores indicating better performance. A total learning score therefore ranges from 0 to 36 and a delayed memory score of 0 to 12, with higher scores reflecting better performance.
Executive Function | Baseline and 12 Weeks
  Executive Function will be assessed using a mean-rank score comprised of the following subtests. The Trail Making Test assesses complex attention, with scores ranging from 10-300 seconds and higher scores reflecting worse performance. The Digit Span task assesses working memory with scores ranging from 0 to 30 and higher scores reflecting better performance. The Digit Symbol Substitution Test assesses visual psychomotor sequencing with scores ranging from 0 to 133 and higher scores reflecting better performance. The Controlled Oral Word Association test assesses verbal flexibility and phonemic fluency over 3, 1-minute time periods, with higher scores reflecting better performance. The Animal Naming Test assesses semantic fluency over 1-minute, with higher scores reflecting better performance. The Stroop Test assess inhibitory control, with higher scores reflecting better performance. The Ruff 2&7 Test assesses psychomotor vigilance, with higher scores reflecting better performance.

SECONDARY OUTCOMES:
Metabolic Flexibility | Baseline and 12 Weeks
  Metabolic flexibility and function will be assessed using a mean-rank, global score comprised of the following biomarkers. Metabolic measures will include Lipids, triglycerides, glucose, insulin, insulin-like growth factor, HbA1c, non-esterified fatty acids, total ketone bodies, brain derived neurotrophic factor, beta-hydroxybutyrate, lactate, amino acids, plasma kynurenine, kynurenic acid, tryptophan, non-esterified fatty acids, and acylcarnitines. All individual biomarkers will be ranked at pre and post treatment before being combined into a mean-rank, global score.
Inflammatory Function | Baseline and 12 Weeks
  Inflammatory function will be assessed using a mean-rank, global score comprised of the following biomarkers. Inflammatory markers will include interleukin6 (IL-6), tumor necrosis factor (TNF)-alpha, high sensitivity C reactive protein (CRP), IL-1β, IL-8, IL-10, myostatin, and glial fibrillary acidic protein (GFAP). All individual biomarkers will be ranked at pre and post treatment before being combined into a mean-rank, global score.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J Smith, PhD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
We will submit de-identified study data to a public database in accordance with the NIH data sharing policy. Datasets will be prepared and submitted to the appropriate program officer no later than 3 years after all patient follow up is complete or 2 years after main manuscript publication of study results (whichever comes first). Dr. Smith will also include documentation and key study documents such as protocol, electronic case report forms, manuals of procedures, and applicable training materials to enable the use of prepared data sets by outside investigators. Data sets and associated documentation will be provided in the preferred electronic format. The prepared and submitted data set will include at minimum baseline, interim visit, procedural and intervention based data, and outcomes data.
Supporting Information: Study Protocol

DOCUMENTS (1):
  • Informed Consent Form (2024-05-29): https://cdn.clinicaltrials.gov/large-docs/16/NCT05997316/ICF_000.pdf